CLINICAL TRIAL: NCT07037706
Title: Use of Macrolides in Acute Chest Syndrome: A Multicenter Retrospective Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0063_REANIMATION
Record Dates: First submitted 2025-06-11; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome; Glucose-6-Phosphate Dehydrogenase Deficiency; Anti-Bacterial Agents; Macrolides
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at whether using macrolide antibiotics is helpful and safe in treating acute chest syndrome, a serious complication in people with sickle cell disease. It reviews past cases from three hospitals where patients were treated in intensive care. The goal is to understand if macrolides make a difference, what germs are involved, how useful lab tests are, and how well patients tolerate these antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old).
* Diagnosis of acute chest syndrome (ACS).
* Hospitalized in an intensive care unit (ICU).
* Microbiological sampling performed (e.g., multiplex PCR, sputum culture [ECBC], and/or Legionella urinary antigen test).
* Received empiric antibiotic therapy including a macrolide.

Exclusion Criteria:

* Minor patient (<18 years old).
* Acute chest syndrome not requiring ICU admission.
* Acute chest syndrome without any attempt at microbiological documentation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 and older) with sickle cell disease who were diagnosed with acute chest syndrome (ACS) and required hospitalization in an intensive care unit (ICU). All selected patients must have received an empiric antibiotic treatment including a macrolide and undergone microbiological sampling (such as PCR multiplex, sputum culture, or urinary antigen testing for Legionella). Participants will be identified retrospectively from medical records across the three participating hospital centers over the study period.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation (in days) among patients with ACS treated with empiric macrolides | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France